CLINICAL TRIAL: NCT01687998
Title: Assessment of Clinical Effects of Cholesteryl Ester Transfer Protein Inhibition With Evacetrapib in Patients at a High-Risk for Vascular Outcomes
Brief Title: A Study of Evacetrapib in High-Risk Vascular Disease
Acronym: ACCELERATE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study termination due to insufficient efficacy.
Sponsor: Eli Lilly and Company (Industry)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11949; I1V-MC-EIAN (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-09-12; First posted 2012-09-19 (Estimated); Results first posted 2018-05-16 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-09

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — evacetrapib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Evacetrapib (Experimental): Evacetrapib 130 mg tablet, administered orally once daily for up to 4 years. Participants will also receive standard of care for high-risk vascular disease (HRVD).
  Interventions: Drug: Evacetrapib
- Placebo (Placebo Comparator): Placebo, tablet administered orally once daily for up to 4 years. Participants will also receive standard of care for HRVD.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Evacetrapib — Administered Orally
  Other Names: LY2484595
  Arms: Evacetrapib
Drug: Placebo — Administered Orally
  Arms: Placebo

SUMMARY:
The purpose of the ACCELERATE study is to evaluate the efficacy and safety of evacetrapib in participants with high-risk vascular disease (HRVD).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of high risk vascular disease (HRVD) (that is, meet at least one of the disease diagnostic criteria of: 1)History of acute coronary syndrome (ACS) (that is, ≥30 days through 365 days after discharge for ACS) 2)cerebrovascular atherosclerotic disease 3)peripheral arterial disease 4)diabetes mellitus with documented coronary artery disease and are clinically stable (as judged by the responsible physician).
* Must be treated with a statin for at least 30 days prior to screening. If not treated with a statin must have documented statin intolerance, or contraindication to statin
* Have a screening high-density lipoprotein cholesterol (HDL-C) ≤80 milligram per deciliter (mg/dL) (≤2.1 millimole per liter [mmol/L])
* Have screening triglycerides (TG) ≤400 mg/dL (≤4.5 mmol/L)
* Meet 1 of the following criteria:

  * screening low-density lipoprotein cholesterol (LDL-C) no more than 10 mg/dL (0.3 mmol/L) above the target chosen by the investigator (either LDL-C <100 mg/dL [<2.6 mmol/L] or LDL-C <70 mg/dL [<1.8 mmol/L]), OR
  * if LDL-C is greater than target, the participant must be on maximum tolerated statin dose (for at least 30 days), have documented statin intolerance, or contraindication to statin

Exclusion Criteria:

* Are currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an investigational product or non-approved use of a drug or device, or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Have previously completed or withdrawn from this study, or withdrawn from any other study investigating evacetrapib
* Female participants who are known to be pregnant or breastfeeding
* Women of child-bearing potential only, who test positive for pregnancy between screening and randomization, or who do not agree to use a reliable method of birth control during the study
* History of transient ischemic attack (TIA) or ischemic stroke <30 days and ACS <30 days
* Any reading of systolic blood pressure ≥180 millimeter of mercury (mm Hg) or diastolic blood pressure ≥110 mm Hg at screening or randomization
* History of hemorrhagic stroke or intracranial hemorrhage
* New York Heart Association class III or IV congestive heart failure
* Serum creatinine >2.2 mg/dL (>194.5 micromole per liter [μmol/L]) at screening
* Clinically active liver disease. Participants are not excluded due to Gilbert's Syndrome or a history of cholelithiasis/cholecystectomy
* History of malignancy within the preceding 3 years prior to screening
* Known malabsorption syndrome with the exception of lactose intolerance
* Participants with a known history of primary or secondary hyperaldosteronism
* Participants with a history of intolerance/hypersensitivity to cholesterol ester transfer protein (CETP) inhibitors
* Any clinically significant medical condition that according to the investigator could interfere with participation in the study
* Participants whose life expectancy is anticipated to be less than 4 years
* Unable or unwilling to comply with study requirements, or deemed by the investigator to be unfit for the study
* Have a history of drug, alcohol, or substance abuse within the past 6 months, as assessed by the investigator
* Concurrent or anticipated need for treatment with niacin >250 mg/day or for chronic administration of drugs on the exclusion list
* Previous exposure to the CETP inhibitors dalcetrapib or evacetrapib within the last 3 months or anacetrapib within the last 12 months
* Any planned coronary angiography or coronary revascularization procedure. If angiography or revascularization is planned, participants may be screened and enrolled after all such planned procedures are completed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12092 (Actual)
Dates: Start 2012-10; Primary Completion 2016-03 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (441):
- United States (176):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Birmingham, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Huntsville, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mobile, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cottonwood, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Glendale, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tucson, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Smith, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Little Rock, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Escondido, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fresno, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lomita, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Long Beach, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mission Viejo, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Rosa, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stockton, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Thousand Oaks, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Torrance, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Colorado Springs, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Golden, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bridgeport, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Waterbury, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aventura, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boynton Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brandon, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Clearwater, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fleming Island, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gainesville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Inverness, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jupiter, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lakeland, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Largo, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Margate, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Melbourne, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miami Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Naples, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ocala, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orlando, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Panama City, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pembroke Pines, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pensacola, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ponte Vedra, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Port Charlotte, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Safety Harbor, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tallahassee, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wellington, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Covington, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cumming, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tucker, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Arlington Heights, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aurora, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bannockburn, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jerseyville, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rock Island, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Anderson, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brownsburg, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Elkhart, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Wayne, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hammond, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Waterloo, Iowa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hutchinson, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Overland Park, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lexington, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Louisville, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baton Rouge, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Covington, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lake Charles, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Auburn, Maine
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bangor, Maine
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbia, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lutherville, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salisbury, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Haverhill, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyannis, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Natick, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Springfield, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cadillac, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lansing, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marquette, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Midland, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Novi, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Petoskey, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pontiac, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saginaw, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Minneapolis, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Cloud, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Paul, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbia, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Springfield, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Great Falls, Montana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Omaha, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bridgewater, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Elizabeth, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Elmer, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Haddon Heights, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mine Hill, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ridgewood, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sewell, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Somerset, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Teaneck, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toms River, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albany, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kingston, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poughkeepsie, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saratoga Springs, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Southampton, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Troy, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Westfield, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Williamsville, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Asheville, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cary, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chapel Hill, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Elizabeth City, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greensboro, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hickory, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lenoir, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wilmington, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beachwood, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Canton, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cleveland, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mansfield, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sandusky, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toledo, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zanesville, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oklahoma City, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tulsa, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portland, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beaver, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bethlehem, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Camp Hill, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Danville, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hershey, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Port Matilda, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pottstown, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Red Lion, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wilkes-Barre, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cumberland, Rhode Island
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbia, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greenville, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greer, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rapid City, South Dakota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greeneville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Knoxville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tullahoma, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Corpus Christi, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kerrville, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kingwood, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tomball, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bountiful, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Murray, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salt Lake City, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charlottesville, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Danville, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Falls Church, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Harrisonburg, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lynchburg, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Roanoke, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bellevue, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tacoma, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Huntington, West Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Green Bay, Wisconsin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madison, Wisconsin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milwaukee, Wisconsin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oregon, Wisconsin
- Argentina (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Belgrano
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Coronel Suárez
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Córdoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Luis
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Miguel de Tucumán
- Australia (12):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Camperdown, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wollongong, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Herston, Queensland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milton, Queensland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Southport, Queensland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Woodville, South Australia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Launceston, Tasmania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Box Hill, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Geelong, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heidelberg, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Melbourne, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Windsor, Victoria
- Austria (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Feldkirch
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Graz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Innsbruck
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vienna
- Belgium (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Antwerp
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brussels
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Huy
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Merksem
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tienen
- Brazil (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fortaleza
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rio de Janeiro
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., São Paulo
- Bulgaria (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gabrovo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pazardzhik
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pleven
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Plovdiv
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Smolyan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sofia
- Canada (21):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kelowna, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mount Pearl, Newfoundland and Labrador
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cambridge, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greater Sudbury, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamilton, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mississauga, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oshawa, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sarnia, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Thunder Bay, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toronto, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brossard, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicoutimi, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gatineau, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greenfield Park, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Joilette, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Longueuil, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montreal, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint-Georges, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint-Jérôme, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint-Lambert, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sainte-Foy, Quebec
- China (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beijing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Changsha
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guangzhou
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Harbin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shanghai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shenyang
- Czechia (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Český Krumlov
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hodonín
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mariánské Lázně
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pardubice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Písek
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prague
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Příbram
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Teplice
- Denmark (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aalborg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ballerup Municipality
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Copenhagen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vejle
- Estonia (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tallinn
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Viljandi
- France (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bordeaux
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dijon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Le Coudray
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pessac
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Strasbourg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toulouse
- Germany (15):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Altenburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bad Krozingen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bielefeld
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dortmund
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dresden
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Frankfurt
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heidelberg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kassel
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mainz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mönchengladbach
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stuttgart
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tübingen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warendorf
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wiesbaden
- Hong Kong (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Central
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hong Kong
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shatin
- Hungary (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Békéscsaba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Budapest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Debrecen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Esztergom
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hódmezővásárhely
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kalocsa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Komárom
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orosháza
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szekszárd
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zalaegerszeg
- Israel (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Haifa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jerusalem
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nazareth
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rehovot
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Safed
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tel Aviv
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tel Litwinsky
- Italy (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bologna
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Castelfranco Veneto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chieti Scalo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Napoli
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Novara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Parma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Piacenza
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Daniele del Friuli
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sessa Aurunca
- Japan (18):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aichi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ehime
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gunma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyōgo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ibaraki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ishikawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kumamoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kyoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Okinawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saitama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shizuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokushima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yamaguchi
- Lithuania (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kaunas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Klaipėda
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vilnius
- Mexico (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aguascalientes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chihuahua City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cul Sinaloa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Huixquilucan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Querétaro
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Luis Potosí City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampico
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tijuana
- Netherlands (18):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., 's-Hertogenbosch
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Amersfoort
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Amsterdam
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beverwijk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Delft
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Den Helder
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Deventer
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Drachten
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heerlen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hilversum
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hoogeveen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hoorn
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leiden
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tilburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Venlo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Waalwijk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zaandam
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zwijndrecht
- New Zealand (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Addington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Grafton
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamilton West
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Newtown
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tauranga
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Westlake
- Poland (12):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bydgoszcz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gdansk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Katowice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Krakow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kutno
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lodz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oława
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Puławy
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Skierniewice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sobótka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wroclaw
- Puerto Rico (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ponce
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Trujillo Alto
- Romania (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brăila
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buzău
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Focşani
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oradea
- Russia (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Arkhangelsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kemerovo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Smolensk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tomsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yaroslavl
- Slovakia (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bardejov
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bratislava
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kráľovský Chlmec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nitra
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prešov
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Žilina
- South Africa (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alberton
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bellville
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bloemfontein
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Goodwood
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Johannesburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kuilsriver
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Newlands West
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Parktown West
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Worcester
- South Korea (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Anyang
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Busan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daejeon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gangwon-Do
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Goyang
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gwangju
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jungbuk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
- Spain (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ciudad Real
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Córdoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., L'Hospitalet de Llobregat
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Málaga
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palma de Mallorca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pamplona
- Sweden (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lund
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Malmo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Östersund
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stockholm
- Switzerland (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lugano
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zurich
- Taiwan (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kaohsiung City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kuei Shan Hsiang
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taichung
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei
- Turkey (Türkiye) (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ankara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Konya
- Ukraine (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kyiv
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lutsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poltava
- United Kingdom (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Stephen, Cornwall
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Welwyn Garden City, Hertfordshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barnet, Herts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stevenage, Herts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tooting, London
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wellingborough, Northants
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dudley, West Midlands
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bath
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Frome

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Puri R, Nissen SE, Arsenault BJ, St John J, Riesmeyer JS, Ruotolo G, McErlean E, Menon V, Cho L, Wolski K, Lincoff AM, Nicholls SJ. Effect of C-Reactive Protein on Lipoprotein(a)-Associated Cardiovascular Risk in Optimally Treated Patients With High-Risk Vascular Disease: A Prespecified Secondary Analysis of the ACCELERATE Trial. JAMA Cardiol. 2020 Oct 1;5(10):1136-1143. doi: 10.1001/jamacardio.2020.2413. PMID 32639518
- [Derived] Menon V, Kumar A, Patel DR, John JS, Wolski KE, McErlean E, Riesmeyer JS, Weerakkody G, Ruotolo G, Cremer PC, Nicholls SJ, Lincoff AM, Nissen SE. Impact of Baseline Glycemic Control on Residual Cardiovascular Risk in Patients With Diabetes Mellitus and High-Risk Vascular Disease Treated With Statin Therapy. J Am Heart Assoc. 2020 Jan 7;9(1):e014328. doi: 10.1161/JAHA.119.014328. Epub 2019 Dec 19. PMID 31852422
- [Derived] Kumar A, Patel DR, Brennan DM, Wolski KE, Lincoff AM, Ruotolo G, McErlean E, Weerakkody G, Riesmeyer JS, Nicholls SJ, Nissen SE, Menon V. Plasma Aldosterone Levels Are Not Associated With Cardiovascular Events Among Patients With High-Risk Vascular Disease: Insights From the ACCELERATE Trial. J Am Heart Assoc. 2019 Dec 3;8(23):e013790. doi: 10.1161/JAHA.119.013790. Epub 2019 Nov 22. PMID 31752637
- [Derived] Lincoff AM, Nicholls SJ, Riesmeyer JS, Barter PJ, Brewer HB, Fox KAA, Gibson CM, Granger C, Menon V, Montalescot G, Rader D, Tall AR, McErlean E, Wolski K, Ruotolo G, Vangerow B, Weerakkody G, Goodman SG, Conde D, McGuire DK, Nicolau JC, Leiva-Pons JL, Pesant Y, Li W, Kandath D, Kouz S, Tahirkheli N, Mason D, Nissen SE; ACCELERATE Investigators. Evacetrapib and Cardiovascular Outcomes in High-Risk Vascular Disease. N Engl J Med. 2017 May 18;376(20):1933-1942. doi: 10.1056/NEJMoa1609581. PMID 28514624

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Non-Completers: Participants "Known to be Alive at Study End" is a subset of those who did not withdraw consent and later found to be alive from public sources. "Lost to follow-up" is a subset of those who did not withdraw consent for whom study end vital status could not be ascertained.
Groups:
- Evacetrapib: Evacetrapib 130 milligram (mg) tablet, administered orally once daily for up to 4 years. Participants will also receive standard of care for high-risk vascular disease (HRVD).
Period: Overall Study
Arm/Group | Evacetrapib | Placebo
Started | 6038 | 6054
Received at Least One Dose of Study Drug | 6036 | 6052
Completed | 5926 | 5934
Not Completed | 112 | 120
Not completed — Withdrawal by Subject | 49 | 51
Not completed — Known to be Alive at Study End | 54 | 62
Not completed — Lost to Follow-up | 9 | 7

BASELINE CHARACTERISTICS:
Groups:
- Evacetrapib: Evacetrapib 130 mg tablet, administered orally once daily for up to 4 years. Participants received standard of care for HRVD.
- Placebo: Placebo, tablet administered orally once daily for up to 4 years. Participants received standard of care for HRVD.
- Total: Total of all reporting groups
Arm/Group | Evacetrapib | Placebo | Total
Number analyzed (Participants) | 6038 | 6054 | 12092
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.791 (9.3849) | 64.994 (9.4591) | 64.892 (9.4223)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1390 | 1394 | 2784
  Male | 4648 | 4660 | 9308
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 500 | 522 | 1022
  Not Hispanic or Latino | 5394 | 5386 | 10780
  Unknown or Not Reported | 144 | 146 | 290
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 243 | 226 | 469
  Asian | 650 | 640 | 1290
  Native Hawaiian or Other Pacific Islander | 6 | 5 | 11
  Black or African American | 141 | 153 | 294
  White | 4933 | 4971 | 9904
  More than one race | 35 | 26 | 61
  Unknown or Not Reported | 30 | 33 | 63
Region of Enrollment [Count of Participants; unit: Participants]
  Russia | 85 | 82 | 167
  Hong Kong | 24 | 28 | 52
  United States | 2235 | 2240 | 4475
  Netherlands | 171 | 169 | 340
  Austria | 34 | 34 | 68
  Sweden | 33 | 33 | 66
  China | 224 | 221 | 445
  South Korea | 87 | 94 | 181
  Poland | 243 | 240 | 483
  Brazil | 54 | 56 | 110
  Slovakia | 116 | 117 | 233
  France | 45 | 52 | 97
  Bulgaria | 113 | 118 | 231
  Lithuania | 13 | 15 | 28
  Argentina | 89 | 91 | 180
  Romania | 64 | 66 | 130
  Hungary | 118 | 115 | 233
  Japan | 205 | 202 | 407
  Ukraine | 67 | 66 | 133
  United Kingdom | 58 | 58 | 116
  Switzerland | 15 | 14 | 29
  Spain | 65 | 66 | 131
  New Zealand | 63 | 64 | 127
  Canada | 626 | 619 | 1245
  Czechia | 187 | 185 | 372
  Turkey | 1 | 2 | 3
  Belgium | 42 | 42 | 84
  Taiwan | 52 | 53 | 105
  Denmark | 95 | 100 | 195
  Italy | 43 | 40 | 83
  Mexico | 235 | 231 | 466
  South Africa | 77 | 76 | 153
  Israel | 72 | 74 | 146
  Australia | 159 | 160 | 319
  Germany | 198 | 202 | 400
  Estonia | 30 | 29 | 59

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Composite Primary Endpoint of Cardiovascular (CV) Death, Myocardial Infarction (MI), Stroke, Coronary Revascularization, or Hospitalization for Unstable Angina (UA)
Description: For component endpoints, the number of participants includes those experiencing fatal events and account for all occurrences regardless of whether or not another component event occurred previously.
Time Frame: Baseline to Study Completion (Up to 4 years)
Population: All randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Evacetrapib | Placebo
Number analyzed (Participants) | 6038 | 6054
Participants | 779 | 776
Statistical Analysis 1: Comparison: Evacetrapib vs Placebo; Primary Endpoint: Time to First Occurrence of the Composite Primary Endpoint of Cardiovascular (CV) Death, Myocardial Infarction (MI), Stroke, Coronary Revascularization, or Hospitalization for Unstable Angina (UA); Test type: Superiority or Other; p = 0.9054, Regression, Cox; Hazard Ratio (HR) = 1.006, 95% CI 2-sided [0.911 to 1.111]

2. Secondary Outcome: Mean Percent Change From Baseline to 3 Months in Low-Density (LDL-C) and High-Density Lipoprotein Cholesterol (HDL-C) Levels
Time Frame: Baseline, 3 Months
Population: All randomized participants with evaluable LDL-C and HDL-C levels.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Evacetrapib | Placebo
Number analyzed (Participants) | 6038 | 6054
percent
  LDL-C: number analyzed (Participants) | 5760 | 5786
  LDL-C | -31.12 (27.583) | 5.99 (29.007)
  HDL-C: number analyzed (Participants) | 5760 | 5788
  HDL-C | 133.18 (57.204) | 1.63 (17.455)
Statistical Analysis 1: Comparison: Evacetrapib vs Placebo; LDL-C; Test type: Superiority or Other; p < 0.0001, ANOVA; Mean Difference (Final Values) = -37.11, 95% CI 2-sided [-38.15 to -36.08]
Statistical Analysis 2: Comparison: Evacetrapib vs Placebo; HDL-C; Test type: Superiority or Other; p < 0.0001, ANOVA; Mean Difference (Final Values) = 131.55, 95% CI 2-sided [130.01 to 133.09]

3. Secondary Outcome: Number of Participants With Composite Endpoint of All-Cause Mortality, MI, Stroke, Coronary Revascularization, or Hospitalization for UA
Description: as for outcome 1
Time Frame: Baseline through End of Study (Up to 4 years)
Population: All randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Evacetrapib | Placebo
Number analyzed (Participants) | 6038 | 6054
Participants | 857 | 867
Statistical Analysis 1: Comparison: Evacetrapib vs Placebo; Time to First Occurrence of the Composite Endpoint of All-Cause Mortality, MI, Stroke, Coronary Revascularization, or Hospitalization for UA; Test type: Superiority or Other; p = 0.8463, Regression, Cox; Hazard Ratio (HR) = 0.991, 95% CI 2-sided [0.901 to 1.089]

4. Secondary Outcome: Number of Participants With Composite Endpoint of CV Death, MI, or Coronary Revascularization
Description: as for outcome 1
Time Frame: Baseline through End of Study (Up to 4 years)
Population: All randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Evacetrapib | Placebo
Number analyzed (Participants) | 6038 | 6054
Participants | 690 | 691
Statistical Analysis 1: Comparison: Evacetrapib vs Placebo; Time to First Occurrence of the Composite Endpoint of CV Death, MI, or Coronary Revascularization; Test type: Superiority or Other; p = 0.9874, Regression, Cox; Hazard Ratio (HR) = 1.001, 95% CI 2-sided [0.901 to 1.112]

5. Secondary Outcome: Number of Participants With Composite Endpoint of CV Death, MI, Stroke, or Hospitalization for UA
Description: as for outcome 1
Time Frame: Baseline through End of Study (Up to 4 years)
Population: All randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Evacetrapib | Placebo
Number analyzed (Participants) | 6038 | 6054
Participants | 571 | 570
Statistical Analysis 1: Comparison: Evacetrapib vs Placebo; Time to First Occurrence of the Composite Endpoint of CV Death, MI, Stroke, or Hospitalization for UA; Test type: Superiority or Other; p = 0.9574, Regression, Cox; Hazard Ratio (HR) = 1.003, 95% CI 2-sided [0.893 to 1.127]

6. Secondary Outcome: Number of Participants With Triple Composite Endpoint of CV Death, MI, or Stroke
Description: as for outcome 1
Time Frame: Baseline through End of Study (Up to 4 years)
Population: All randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Evacetrapib | Placebo
Number analyzed (Participants) | 6038 | 6054
Participants | 437 | 453
Statistical Analysis 1: Comparison: Evacetrapib vs Placebo; Time to First Occurrence of Triple Composite Endpoint of CV Death, MI, or Stroke; Test type: Superiority or Other; p = 0.5917, Regression, Cox; Hazard Ratio (HR) = 0.965, 95% CI 2-sided [0.846 to 1.100]

ADVERSE EVENTS:
Description: All randomized participants who received at least one dose of study drug. 4 participants were randomized but never took drug and were not in the safety population. 2 females were assigned to evacetrapib and 2 males were assigned to placebo.
Arm/Group | Evacetrapib | Placebo
Serious Adverse Events (participants affected / at risk) | 2306/6036 | 2341/6052
Other Adverse Events (participants affected / at risk) | 2659/6036 | 2529/6052
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Evacetrapib (N=6036) | Placebo (N=6052)
Anaemia (Blood and lymphatic system disorders) | 30 (31) | 38 (46)
Aplastic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Cytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (4) | 0 (0)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1) | 5 (6)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (2) | 5 (5)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 4 (4)
Lymphadenitis (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Microcytic anaemia (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Pancytopenia (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Pernicious anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Spontaneous haemorrhage (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Acute coronary syndrome (Cardiac disorders) | 9 (9) | 4 (4)
Acute myocardial infarction (Cardiac disorders) | 146 (168) | 137 (149)
Adams-stokes syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 102 (113) | 98 (103)
Angina unstable (Cardiac disorders) | 298 (389) | 289 (363)
Aortic valve disease (Cardiac disorders) | 4 (4) | 1 (1)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 2 (2)
Aortic valve sclerosis (Cardiac disorders) | 0 (0) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 7 (7) | 6 (8)
Arrhythmia (Cardiac disorders) | 5 (5) | 3 (3)
Arteriosclerosis coronary artery (Cardiac disorders) | 2 (3) | 1 (1)
Arteriospasm coronary (Cardiac disorders) | 1 (1) | 1 (2)
Atrial fibrillation (Cardiac disorders) | 86 (109) | 78 (94)
Atrial flutter (Cardiac disorders) | 25 (27) | 16 (18)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Atrial thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block (Cardiac disorders) | 5 (5) | 3 (3)
Atrioventricular block complete (Cardiac disorders) | 8 (8) | 6 (6)
Atrioventricular block second degree (Cardiac disorders) | 6 (6) | 1 (1)
Bradyarrhythmia (Cardiac disorders) | 0 (0) | 5 (5)
Bradycardia (Cardiac disorders) | 8 (8) | 11 (11)
Cardiac arrest (Cardiac disorders) | 17 (18) | 30 (32)
Cardiac discomfort (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 67 (79) | 63 (78)
Cardiac failure acute (Cardiac disorders) | 11 (13) | 9 (9)
Cardiac failure chronic (Cardiac disorders) | 7 (7) | 10 (12)
Cardiac failure congestive (Cardiac disorders) | 95 (134) | 103 (138)
Cardiac tamponade (Cardiac disorders) | 2 (2) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 5 (5) | 6 (7)
Cardiogenic shock (Cardiac disorders) | 8 (8) | 7 (7)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 5 (5)
Cardiopulmonary failure (Cardiac disorders) | 3 (3) | 0 (0)
Cardiorenal syndrome (Cardiac disorders) | 2 (2) | 1 (1)
Cardiovascular insufficiency (Cardiac disorders) | 1 (1) | 0 (0)
Chronotropic incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Conduction disorder (Cardiac disorders) | 4 (4) | 1 (1)
Congestive cardiomyopathy (Cardiac disorders) | 1 (1) | 2 (2)
Coronary artery disease (Cardiac disorders) | 37 (40) | 44 (45)
Coronary artery dissection (Cardiac disorders) | 2 (2) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 3 (3) | 6 (6)
Coronary artery stenosis (Cardiac disorders) | 7 (7) | 6 (7)
Diastolic dysfunction (Cardiac disorders) | 2 (2) | 1 (1)
Dressler's syndrome (Cardiac disorders) | 1 (1) | 2 (2)
Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Hypertensive heart disease (Cardiac disorders) | 1 (1) | 0 (0)
Intracardiac thrombus (Cardiac disorders) | 1 (1) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 7 (7) | 10 (11)
Left ventricular dysfunction (Cardiac disorders) | 5 (6) | 3 (4)
Left ventricular failure (Cardiac disorders) | 0 (0) | 4 (4)
Microvascular coronary artery disease (Cardiac disorders) | 0 (0) | 2 (2)
Mitral valve incompetence (Cardiac disorders) | 3 (4) | 4 (6)
Mitral valve stenosis (Cardiac disorders) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 82 (88) | 100 (107)
Myocardial ischaemia (Cardiac disorders) | 15 (16) | 9 (9)
Myocardial rupture (Cardiac disorders) | 1 (1) | 0 (0)
Nodal rhythm (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 6 (6) | 2 (2)
Pericardial effusion (Cardiac disorders) | 1 (1) | 2 (2)
Pericardial haemorrhage (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 5 (5) | 2 (2)
Postinfarction angina (Cardiac disorders) | 0 (0) | 1 (1)
Prinzmetal angina (Cardiac disorders) | 0 (0) | 2 (2)
Right ventricular failure (Cardiac disorders) | 3 (3) | 2 (2)
Sinus arrest (Cardiac disorders) | 2 (2) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 3 (3)
Sinus node dysfunction (Cardiac disorders) | 12 (12) | 9 (9)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 3 (3) | 6 (6)
Systolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Ventricle rupture (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 4 (4) | 2 (2)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 4 (4)
Ventricular fibrillation (Cardiac disorders) | 7 (7) | 10 (10)
Ventricular hypokinesia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 16 (21) | 24 (24)
Wolff-parkinson-white syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Arteriovenous malformation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Atrial septal defect (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Dermoid cyst (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 2/4658 (2)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Leukodystrophy (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Phimosis (Congenital, familial and genetic disorders) | 0 (0) | 1/4658 (1)
Conductive deafness (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Deafness neurosensory (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Meniere's disease (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Otosclerosis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 7 (7) | 15 (15)
Vertigo positional (Ear and labyrinth disorders) | 5 (5) | 2 (2)
Autoimmune thyroiditis (Endocrine disorders) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 1 (1) | 3 (3)
Hyperparathyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hyperparathyroidism primary (Endocrine disorders) | 0 (0) | 1 (1)
Age-related macular degeneration (Eye disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 15 (19) | 14 (14)
Cataract nuclear (Eye disorders) | 2 (2) | 2 (3)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Diabetic retinopathy (Eye disorders) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Ectropion (Eye disorders) | 0 (0) | 1 (1)
Entropion (Eye disorders) | 1 (1) | 0 (0)
Eye haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Eyelid ptosis (Eye disorders) | 3 (3) | 1 (1)
Glaucoma (Eye disorders) | 3 (3) | 2 (3)
Idiopathic orbital inflammation (Eye disorders) | 1 (1) | 0 (0)
Iridocyclitis (Eye disorders) | 1 (1) | 0 (0)
Iritis (Eye disorders) | 1 (1) | 0 (0)
Keratitis (Eye disorders) | 1 (1) | 0 (0)
Keratopathy (Eye disorders) | 1 (1) | 0 (0)
Lens dislocation (Eye disorders) | 0 (0) | 1 (1)
Macular fibrosis (Eye disorders) | 1 (1) | 1 (1)
Open angle glaucoma (Eye disorders) | 0 (0) | 1 (1)
Optic atrophy (Eye disorders) | 1 (1) | 0 (0)
Optic ischaemic neuropathy (Eye disorders) | 0 (0) | 2 (2)
Optic neuropathy (Eye disorders) | 0 (0) | 1 (1)
Retinal artery occlusion (Eye disorders) | 1 (1) | 1 (1)
Retinal detachment (Eye disorders) | 2 (2) | 2 (2)
Retinal haemorrhage (Eye disorders) | 1 (1) | 1 (1)
Retinopathy (Eye disorders) | 0 (0) | 1 (1)
Visual acuity reduced (Eye disorders) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 1 (1)
Abdominal adhesions (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal compartment syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 2 (2) | 3 (3)
Abdominal mass (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 18 (20) | 8 (8)
Abdominal pain upper (Gastrointestinal disorders) | 5 (5) | 7 (7)
Abdominal strangulated hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal wall cyst (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal wall haematoma (Gastrointestinal disorders) | 1 (1) | 1 (1)
Alcoholic pancreatitis (Gastrointestinal disorders) | 0 (0) | 2 (4)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 2 (2)
Chronic gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Coeliac artery stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 5 (5) | 9 (9)
Colitis ischaemic (Gastrointestinal disorders) | 4 (4) | 6 (7)
Colitis microscopic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colonic fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (5) | 8 (8)
Crohn's disease (Gastrointestinal disorders) | 1 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 6 (7) | 4 (4)
Dieulafoy's vascular malformation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diverticulum intestinal (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 5 (5) | 2 (2)
Duodenal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 3 (3) | 3 (3)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 3 (3)
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 (0) | 3 (3)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Enteritis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterovesical fistula (Gastrointestinal disorders) | 1 (1) | 1 (1)
Erosive oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Faecal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 4 (4)
Femoral hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric cyst (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric disorder (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 6 (6) | 7 (7)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastric ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 10 (10) | 10 (10)
Gastritis alcoholic (Gastrointestinal disorders) | 0 (0) | 1 (3)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastrointestinal angiodysplasia haemorrhagic (Gastrointestinal disorders) | 0 (0) | 3 (3)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (2) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 32 (32) | 26 (32)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 13 (13) | 11 (11)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (2)
Glossitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 3 (3) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 3 (3) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 4 (4) | 2 (2)
Heyde's syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 4 (4) | 2 (2)
Ileus (Gastrointestinal disorders) | 5 (5) | 5 (5)
Impaired gastric emptying (Gastrointestinal disorders) | 2 (3) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 15 (15) | 13 (14)
Intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal infarction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 5 (6) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 6 (6)
Intestinal perforation (Gastrointestinal disorders) | 2 (2) | 3 (3)
Intestinal prolapse (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intra-abdominal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Jejunal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Large intestinal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 2 (2) | 2 (2)
Large intestine polyp (Gastrointestinal disorders) | 6 (7) | 11 (12)
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 6 (6) | 4 (4)
Mallory-weiss syndrome (Gastrointestinal disorders) | 0 (0) | 2 (2)
Melaena (Gastrointestinal disorders) | 3 (3) | 3 (3)
Mesenteric vascular insufficiency (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (8) | 6 (6)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oedematous pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal achalasia (Gastrointestinal disorders) | 2 (3) | 0 (0)
Oesophageal oedema (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal spasm (Gastrointestinal disorders) | 0 (0) | 2 (2)
Oesophageal stenosis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Pancreatic mass (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic pseudocyst (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 12 (13) | 10 (11)
Pancreatitis acute (Gastrointestinal disorders) | 10 (10) | 6 (6)
Pancreatitis chronic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis necrotising (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 2 (2)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Peritoneal adhesions (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumoperitoneum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Rectal polyp (Gastrointestinal disorders) | 1 (1) | 2 (2)
Rectal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retroperitoneal effusion (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 2 (2) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (3)
Salivary gland mass (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 11 (12) | 10 (11)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Swollen tongue (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tongue haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tongue oedema (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 3 (3) | 6 (6)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 11 (12) | 10 (10)
Volvulus (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 9 (12) | 7 (7)
Adverse drug reaction (General disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 5 (5) | 9 (9)
Cardiac death (General disorders) | 0 (0) | 5 (5)
Chest discomfort (General disorders) | 7 (7) | 12 (13)
Chest pain (General disorders) | 37 (38) | 34 (42)
Death (General disorders) | 20 (20) | 14 (14)
Device breakage (General disorders) | 0 (0) | 2 (2)
Device dislocation (General disorders) | 4 (5) | 1 (1)
Device end of service (General disorders) | 0 (0) | 1 (1)
Device failure (General disorders) | 2 (2) | 2 (2)
Device inappropriate shock delivery (General disorders) | 1 (1) | 0 (0)
Device malfunction (General disorders) | 1 (1) | 6 (6)
Device material issue (General disorders) | 1 (1) | 1 (1)
Device occlusion (General disorders) | 2 (2) | 0 (0)
Drowning (General disorders) | 0 (0) | 1 (1)
Drug withdrawal syndrome (General disorders) | 1 (1) | 0 (0)
Exercise tolerance decreased (General disorders) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 2 (2) | 1 (1)
General physical health deterioration (General disorders) | 2 (2) | 1 (1)
Generalised oedema (General disorders) | 3 (3) | 0 (0)
Granuloma (General disorders) | 0 (0) | 1 (1)
Hyperthermia (General disorders) | 0 (0) | 2 (2)
Hypertrophy (General disorders) | 1 (1) | 0 (0)
Hypothermia (General disorders) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 2 (2) | 3 (3)
Implant site haematoma (General disorders) | 1 (1) | 0 (0)
Incarcerated hernia (General disorders) | 1 (1) | 3 (4)
Ischaemic ulcer (General disorders) | 0 (0) | 2 (2)
Lead dislodgement (General disorders) | 0 (0) | 2 (2)
Multi-organ failure (General disorders) | 4 (4) | 6 (6)
Necrobiosis (General disorders) | 0 (0) | 1 (1)
Necrosis (General disorders) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 107 (123) | 108 (118)
Oedema (General disorders) | 1 (3) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 3 (3)
Pain (General disorders) | 2 (2) | 0 (0)
Pelvic mass (General disorders) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 1 (1)
Precancerous mucosal lesion (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 4 (4)
Stent-graft endoleak (General disorders) | 0 (0) | 1 (1)
Sudden cardiac death (General disorders) | 16 (16) | 15 (15)
Sudden death (General disorders) | 2 (2) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 4 (4) | 0 (0)
Thrombosis in device (General disorders) | 0 (0) | 1 (1)
Ulcer haemorrhage (General disorders) | 1 (1) | 2 (2)
Vascular stent occlusion (General disorders) | 1 (1) | 2 (2)
Vascular stent restenosis (General disorders) | 6 (6) | 5 (6)
Vascular stent stenosis (General disorders) | 1 (1) | 1 (1)
Vascular stent thrombosis (General disorders) | 0 (0) | 2 (2)
Vessel puncture site haematoma (General disorders) | 0 (0) | 1 (1)
Autoimmune hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 5 (6) | 10 (11)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Biliary tract disorder (Hepatobiliary disorders) | 1 (1) | 2 (2)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 4 (4)
Cholangitis acute (Hepatobiliary disorders) | 1 (1) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 19 (20) | 16 (16)
Cholecystitis acute (Hepatobiliary disorders) | 12 (12) | 15 (16)
Cholecystitis chronic (Hepatobiliary disorders) | 4 (4) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 23 (23) | 22 (23)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Gallbladder disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 2 (2) | 3 (3)
Hepatic lesion (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hepatitis alcoholic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hydrocholecystis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Ischaemic hepatitis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Jaundice (Hepatobiliary disorders) | 0 (0) | 3 (3)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice extrahepatic obstructive (Hepatobiliary disorders) | 1 (1) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 1 (1)
Anaphylactic shock (Immune system disorders) | 1 (1) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Abdominal abscess (Infections and infestations) | 3 (3) | 5 (5)
Abdominal infection (Infections and infestations) | 2 (2) | 0 (0)
Abdominal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Abdominal wall abscess (Infections and infestations) | 1 (1) | 1 (1)
Abdominal wall infection (Infections and infestations) | 1 (2) | 0 (0)
Abscess (Infections and infestations) | 1 (1) | 2 (2)
Abscess limb (Infections and infestations) | 3 (3) | 4 (4)
Abscess neck (Infections and infestations) | 1 (1) | 1 (1)
Abscess of salivary gland (Infections and infestations) | 0 (0) | 1 (1)
Abscess oral (Infections and infestations) | 1 (1) | 1 (1)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 1 (1)
Appendicitis (Infections and infestations) | 9 (9) | 5 (5)
Appendicitis perforated (Infections and infestations) | 1 (1) | 2 (2)
Arteriosclerotic gangrene (Infections and infestations) | 1 (2) | 0 (0)
Arteritis infective (Infections and infestations) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 1 (1) | 1 (1)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 6 (7) | 5 (6)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 3 (3) | 2 (2)
Biliary sepsis (Infections and infestations) | 0 (0) | 1 (1)
Biliary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Breast cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 25 (25) | 18 (18)
Bronchitis viral (Infections and infestations) | 1 (1) | 1 (1)
Bursitis infective (Infections and infestations) | 1 (1) | 3 (3)
Cellulitis (Infections and infestations) | 41 (48) | 42 (45)
Cellulitis staphylococcal (Infections and infestations) | 1 (1) | 2 (2)
Cholangitis infective (Infections and infestations) | 1 (1) | 0 (0)
Cholecystitis infective (Infections and infestations) | 5 (5) | 3 (3)
Chronic sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 8 (10)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile sepsis (Infections and infestations) | 0 (0) | 1 (1)
Colonic abscess (Infections and infestations) | 1 (1) | 1 (1)
Cystitis (Infections and infestations) | 6 (6) | 2 (2)
Device related infection (Infections and infestations) | 1 (1) | 2 (2)
Diabetic foot infection (Infections and infestations) | 1 (1) | 1 (1)
Diabetic gangrene (Infections and infestations) | 2 (2) | 0 (0)
Diverticulitis (Infections and infestations) | 13 (13) | 5 (5)
Endocarditis (Infections and infestations) | 2 (4) | 1 (2)
Endocarditis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis enterococcal (Infections and infestations) | 0 (0) | 1 (1)
Endophthalmitis (Infections and infestations) | 2 (2) | 0 (0)
Enterobacter infection (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal infection (Infections and infestations) | 0 (0) | 2 (2)
Enterococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Epididymitis (Infections and infestations) | 1/4648 (1) | 1/4658 (1)
Erysipelas (Infections and infestations) | 6 (8) | 5 (5)
Escherichia bacteraemia (Infections and infestations) | 2 (2) | 0 (0)
Escherichia infection (Infections and infestations) | 0 (0) | 1 (1)
Escherichia pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 2 (2)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 2 (2)
Extradural abscess (Infections and infestations) | 1 (1) | 1 (1)
Febrile infection (Infections and infestations) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1)
Gallbladder abscess (Infections and infestations) | 0 (0) | 1 (1)
Gallbladder empyema (Infections and infestations) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 7 (7) | 11 (14)
Gastritis viral (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 16 (19) | 16 (16)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 8 (8) | 3 (3)
Giardiasis (Infections and infestations) | 0 (0) | 1 (1)
Graft infection (Infections and infestations) | 2 (2) | 1 (1)
Groin abscess (Infections and infestations) | 0 (0) | 1 (1)
H1n1 influenza (Infections and infestations) | 0 (0) | 1 (1)
Haematoma infection (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis c (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis viral (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 2 (2) | 2 (2)
Implant site cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Implant site infection (Infections and infestations) | 0 (0) | 1 (1)
Incision site infection (Infections and infestations) | 2 (2) | 0 (0)
Infected bite (Infections and infestations) | 1 (1) | 0 (0)
Infected fistula (Infections and infestations) | 0 (0) | 1 (1)
Infected seroma (Infections and infestations) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 4 (4) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Infectious colitis (Infections and infestations) | 1 (1) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 2 (2)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (1) | 3 (4)
Influenza (Infections and infestations) | 11 (11) | 9 (9)
Infusion site cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Infusion site infection (Infections and infestations) | 0 (0) | 1 (1)
Intervertebral discitis (Infections and infestations) | 2 (2) | 0 (0)
Keratitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 1 (1) | 0 (0)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 2 (2) | 4 (5)
Lower respiratory tract infection (Infections and infestations) | 2 (3) | 7 (7)
Lung abscess (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Mastoiditis (Infections and infestations) | 1 (1) | 0 (0)
Mediastinitis (Infections and infestations) | 1 (1) | 0 (0)
Myelitis (Infections and infestations) | 0 (0) | 1 (1)
Nail bed infection (Infections and infestations) | 0 (0) | 1 (1)
Necrotising fasciitis (Infections and infestations) | 1 (1) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Orbital infection (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 13 (15) | 5 (6)
Osteomyelitis acute (Infections and infestations) | 1 (1) | 1 (1)
Osteomyelitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis chronic (Infections and infestations) | 0 (0) | 1 (1)
Parainfluenzae virus infection (Infections and infestations) | 1 (1) | 1 (1)
Parotitis (Infections and infestations) | 0 (0) | 1 (1)
Parvovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Pelvic abscess (Infections and infestations) | 0 (0) | 1 (1)
Penile abscess (Infections and infestations) | 1/4648 (1) | 0 (0)
Perihepatic abscess (Infections and infestations) | 1 (1) | 0 (0)
Periodontitis (Infections and infestations) | 1 (1) | 1 (1)
Perirectal abscess (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 3 (3) | 1 (1)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 2 (2)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Pilonidal cyst (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 115 (128) | 112 (122)
Pneumonia bacterial (Infections and infestations) | 2 (2) | 6 (6)
Pneumonia chlamydial (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia fungal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia influenzal (Infections and infestations) | 2 (3) | 0 (0)
Pneumonia legionella (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia parainfluenzae viral (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 1 (1) | 1 (1)
Post procedural cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
Post procedural sepsis (Infections and infestations) | 1 (1) | 0 (0)
Postoperative abscess (Infections and infestations) | 0 (0) | 2 (2)
Postoperative wound infection (Infections and infestations) | 4 (4) | 6 (6)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 2 (2)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 2 (2)
Pyelonephritis (Infections and infestations) | 7 (7) | 4 (4)
Pyelonephritis acute (Infections and infestations) | 2 (2) | 1 (1)
Pyelonephritis chronic (Infections and infestations) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 2 (2) | 3 (4)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1)
Rhinovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Salmonellosis (Infections and infestations) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 44 (49) | 28 (32)
Septic shock (Infections and infestations) | 10 (10) | 7 (7)
Sialoadenitis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2) | 2 (2)
Sinusitis fungal (Infections and infestations) | 0 (0) | 1 (1)
Skin candida (Infections and infestations) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Spinal cord abscess (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 3 (3)
Staphylococcal infection (Infections and infestations) | 6 (6) | 1 (1)
Staphylococcal mediastinitis (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 2 (2)
Streptococcal bacteraemia (Infections and infestations) | 2 (2) | 3 (3)
Streptococcal sepsis (Infections and infestations) | 2 (2) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 1 (2)
Tooth infection (Infections and infestations) | 1 (1) | 1 (1)
Tracheobronchitis (Infections and infestations) | 3 (3) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 2 (2)
Urinary tract infection (Infections and infestations) | 19 (22) | 32 (36)
Urinary tract infection bacterial (Infections and infestations) | 2 (2) | 1 (1)
Urinary tract infection pseudomonal (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 16 (17) | 14 (14)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 3 (3)
Viral labyrinthitis (Infections and infestations) | 1 (1) | 0 (0)
Wound abscess (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 4 (4) | 7 (8)
Wound infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Wound infection staphylococcal (Infections and infestations) | 2 (2) | 1 (1)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Accident (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Accidental exposure to product (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anastomotic stenosis (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Anastomotic ulcer haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 9 (9) | 5 (5)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Brain contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Cartilage injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Chemical burn of skin (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Chemical injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Colon injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Contrast media reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 4 (4) | 4 (4)
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Crush injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cystitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Extradural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Eye injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 39 (40) | 50 (53)
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 (2) | 6 (6)
Femur fracture (Injury, poisoning and procedural complications) | 6 (6) | 6 (6)
Fibula fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Foot fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Foreign body (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Fractured sacrum (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrointestinal anastomotic complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastrointestinal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Graft thrombosis (Injury, poisoning and procedural complications) | 2 (3) | 3 (3)
Gun shot wound (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Head injury (Injury, poisoning and procedural complications) | 6 (6) | 3 (3)
Heat illness (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 6 (6) | 7 (7)
Humerus fracture (Injury, poisoning and procedural complications) | 3 (3) | 4 (4)
Incisional hernia (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
Injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 5 (6) | 2 (2)
Joint injury (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Laceration (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 4 (6) | 2 (2)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 3 (4)
Muscle contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Nerve root injury lumbar (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Peripheral arterial reocclusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Peripheral artery restenosis (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Poisoning (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Post concussion syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post laminectomy syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural bile leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 4 (4) | 4 (4)
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 5 (6) | 3 (3)
Post procedural stroke (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative fever (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative ileus (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 1 (1) | 2 (3)
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural hypotension (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pubis fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Pulmonary contusion (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Radius fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 5 (5) | 8 (8)
Road traffic accident (Injury, poisoning and procedural complications) | 15 (15) | 15 (15)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Soft tissue injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 3 (3) | 5 (5)
Spinal cord injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Splenic rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sternal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 7 (7) | 7 (7)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Tendon injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 8 (9) | 7 (7)
Thermal burn (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 5 (5) | 4 (4)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 3 (3) | 4 (4)
Traumatic amputation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic liver injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 7 (7) | 7 (7)
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 3 (3) | 2 (3)
Vascular pseudoaneurysm ruptured (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Angiogram (Investigations) | 7 (7) | 7 (7)
Anticoagulation drug level above therapeutic (Investigations) | 2 (2) | 0 (0)
Arteriogram (Investigations) | 1 (1) | 0 (0)
Arteriogram coronary (Investigations) | 16 (16) | 17 (17)
Arteriogram renal (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Biopsy brain (Investigations) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 2 (2)
Blood glucose decreased (Investigations) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 1 (1) | 0 (0)
Blood osmolarity decreased (Investigations) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 1 (1) | 0 (0)
Cardiac function test (Investigations) | 0 (0) | 1 (1)
Cardiac stress test abnormal (Investigations) | 0 (0) | 1 (1)
Cardiovascular evaluation (Investigations) | 1 (1) | 1 (1)
Cardiovascular examination (Investigations) | 0 (0) | 1 (1)
Carotid bruit (Investigations) | 1 (1) | 0 (0)
Catheterisation cardiac (Investigations) | 10 (11) | 14 (15)
Clostridium test positive (Investigations) | 0 (0) | 1 (1)
Colonoscopy (Investigations) | 1 (1) | 1 (1)
Computerised tomogram (Investigations) | 1 (1) | 0 (0)
Computerised tomogram thorax (Investigations) | 1 (1) | 0 (0)
Diagnostic procedure (Investigations) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 5 (5) | 4 (4)
Electrocardiogram abnormal (Investigations) | 0 (0) | 1 (1)
Electrocardiogram qt prolonged (Investigations) | 1 (1) | 0 (0)
Endoscopy gastrointestinal (Investigations) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Heart rate irregular (Investigations) | 1 (1) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 1 (1)
International normalised ratio decreased (Investigations) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0)
Investigation (Investigations) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 2 (2) | 0 (0)
Myocardial necrosis marker increased (Investigations) | 2 (2) | 1 (1)
Oesophagogastroduodenoscopy (Investigations) | 1 (1) | 0 (0)
Peripheral arteriogram (Investigations) | 0 (0) | 1 (1)
Prostatic specific antigen increased (Investigations) | 2/4648 (2) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
Troponin increased (Investigations) | 2 (2) | 2 (2)
Ureteroscopy (Investigations) | 1 (1) | 0 (0)
Vitamin b12 decreased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 15 (15) | 26 (28)
Diabetes mellitus (Metabolism and nutrition disorders) | 11 (11) | 20 (22)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 8 (9) | 14 (15)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 2 (4)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Fluid overload (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Gout (Metabolism and nutrition disorders) | 4 (4) | 6 (6)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 13 (13) | 10 (11)
Hyperkalaemia (Metabolism and nutrition disorders) | 9 (9) | 9 (10)
Hyperosmolar hyperglycaemic state (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 17 (17) | 18 (18)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4) | 7 (7)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 6 (7) | 9 (9)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 5 (5) | 5 (5)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 6 (6) | 6 (6)
Vitamin b12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (8) | 17 (19)
Arthritis (Musculoskeletal and connective tissue disorders) | 9 (10) | 7 (7)
Arthropathy (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 15 (15) | 14 (14)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (4)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 7 (8) | 6 (6)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 6 (6) | 14 (15)
Joint instability (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Kyphosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Ligament laxity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 13 (13) | 23 (24)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 17 (18) | 15 (15)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteitis (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 70 (76) | 66 (75)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (7) | 2 (2)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 6 (6) | 3 (3)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 8 (8) | 3 (3)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 6 (6) | 10 (10)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 (5) | 8 (9)
Spinal pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 5 (5)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Adenosquamous cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Anaplastic astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
B-cell lymphoma stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 17 (17) | 13 (16)
Basosquamous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign neoplasm of adrenal gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign neoplasm of spinal cord (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 3 (3)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 5 (7)
Borderline mucinous tumour of ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 4 (4)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (3)
Bronchial neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (3)
Burkitt's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Buschke-lowenstein's tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Carcinoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carcinoid tumour of the gastrointestinal tract (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/1388 (1) | 0 (0)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (4)
Chronic lymphocytic leukaemia stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 2 (2)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 7 (7)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Colon cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer stage iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0)
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colorectal cancer stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Desmoplastic melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Diffuse large b-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Diffuse large b-cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Diffuse large b-cell lymphoma stage ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Diffuse large b-cell lymphoma stage iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Ewing's sarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Fallopian tube cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1/1394 (1)
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gallbladder adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (5) | 6 (7)
Gastrointestinal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrooesophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gingival cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 3 (4)
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (2)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hodgkin's disease stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Keratinising squamous cell carcinoma of nasopharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Laryngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 7 (8)
Lung adenocarcinoma stage i (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma stage ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma stage iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lung carcinoma cell type unspecified stage ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Lung carcinoma cell type unspecified stage iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung carcinoma cell type unspecified stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 (15) | 13 (13)
Lung squamous cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung squamous cell carcinoma stage i (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung squamous cell carcinoma stage iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lymphocytic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Malignant fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 6 (8)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Mediastinum neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Meningioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (5)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Metastases to salivary gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Myxofibrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Nasal sinus cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Nasopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1/4658 (1)
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neuroendocrine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Non-hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-small cell lung cancer stage iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-small cell lung cancer stage iiia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-small cell lung cancer stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Oesophageal adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (1)
Oesophageal adenocarcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Oral cavity cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oropharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oropharyngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 7 (8)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Papillary cystadenoma lymphomatosum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Phaeochromocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 26/4648 (26) | 28/4658 (28)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1/4658 (1)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3/4648 (3) | 0 (0)
Prostate cancer stage ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/4648 (2) | 1/4658 (1)
Prostate cancer stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1/4658 (1)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/4648 (1) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Renal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 2 (2)
Sinonasal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Spinal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (7) | 1 (1)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (8) | 3 (3)
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Squamous cell carcinoma of the vulva (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Testicular neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/4648 (1) | 0 (0)
Testicular seminoma (pure) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1/4658 (1)
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thymoma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tongue carcinoma stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tonsil cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4)
Transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1/1394 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/1388 (1) | 0 (0)
Uterine neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1/1394 (1)
Acute disseminated encephalomyelitis (Nervous system disorders) | 1 (1) | 0 (0)
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 1 (1)
Autonomic nervous system imbalance (Nervous system disorders) | 0 (0) | 1 (1)
Brain injury (Nervous system disorders) | 1 (1) | 2 (2)
Brain mass (Nervous system disorders) | 0 (0) | 1 (1)
Brain stem stroke (Nervous system disorders) | 1 (1) | 0 (0)
Carotid arteriosclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery disease (Nervous system disorders) | 1 (1) | 4 (4)
Carotid artery occlusion (Nervous system disorders) | 1 (1) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 21 (21) | 39 (42)
Carotid sinus syndrome (Nervous system disorders) | 2 (2) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 2 (2) | 2 (2)
Cerebellar ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebellar syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral arteriosclerosis (Nervous system disorders) | 2 (2) | 1 (1)
Cerebral artery occlusion (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 3 (3) | 3 (3)
Cerebral infarction (Nervous system disorders) | 5 (5) | 4 (4)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 3 (4)
Cerebrovascular accident (Nervous system disorders) | 61 (63) | 62 (65)
Cerebrovascular insufficiency (Nervous system disorders) | 0 (0) | 1 (1)
Cervical myelopathy (Nervous system disorders) | 0 (0) | 1 (1)
Cervical radiculopathy (Nervous system disorders) | 1 (1) | 3 (3)
Cognitive disorder (Nervous system disorders) | 1 (1) | 2 (2)
Complex partial seizures (Nervous system disorders) | 0 (0) | 1 (1)
Complex regional pain syndrome (Nervous system disorders) | 0 (0) | 1 (2)
Dementia (Nervous system disorders) | 3 (4) | 3 (3)
Dementia alzheimer's type (Nervous system disorders) | 3 (3) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 6 (9) | 2 (2)
Dizziness (Nervous system disorders) | 6 (6) | 6 (7)
Embolic cerebral infarction (Nervous system disorders) | 2 (2) | 0 (0)
Embolic stroke (Nervous system disorders) | 1 (1) | 1 (1)
Encephalopathy (Nervous system disorders) | 4 (4) | 4 (5)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Essential tremor (Nervous system disorders) | 1 (1) | 0 (0)
Guillain-barre syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 3 (3) | 5 (5)
Haemorrhagic transformation stroke (Nervous system disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 7 (7) | 2 (2)
Hemiparesis (Nervous system disorders) | 3 (3) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 2 (2)
Hypoglycaemic coma (Nervous system disorders) | 0 (0) | 1 (1)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 (1) | 2 (2)
Intraventricular haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 25 (25) | 18 (19)
Lacunar infarction (Nervous system disorders) | 2 (2) | 2 (2)
Loss of consciousness (Nervous system disorders) | 1 (1) | 2 (2)
Lumbar radiculopathy (Nervous system disorders) | 3 (3) | 2 (2)
Lumbosacral radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 3 (3) | 5 (5)
Migraine (Nervous system disorders) | 5 (5) | 0 (0)
Moyamoya disease (Nervous system disorders) | 0 (0) | 1 (1)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 1 (2)
Myelitis transverse (Nervous system disorders) | 1 (1) | 0 (0)
Myoclonus (Nervous system disorders) | 0 (0) | 1 (1)
Nerve compression (Nervous system disorders) | 1 (1) | 1 (1)
Nerve root compression (Nervous system disorders) | 0 (0) | 1 (1)
Nervous system disorder (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 1 (1)
Normal pressure hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Parkinson's disease (Nervous system disorders) | 1 (1) | 0 (0)
Partial seizures (Nervous system disorders) | 0 (0) | 3 (3)
Peroneal nerve palsy (Nervous system disorders) | 1 (1) | 1 (1)
Polyneuropathy (Nervous system disorders) | 0 (0) | 2 (2)
Post herpetic neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Postictal paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 8 (9) | 9 (9)
Quadriparesis (Nervous system disorders) | 1 (1) | 1 (1)
Quadriplegia (Nervous system disorders) | 1 (1) | 0 (0)
Radicular syndrome (Nervous system disorders) | 0 (0) | 2 (2)
Radiculopathy (Nervous system disorders) | 2 (2) | 2 (8)
Restless legs syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 6 (6) | 4 (4)
Seizure (Nervous system disorders) | 7 (7) | 6 (6)
Spinal claudication (Nervous system disorders) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (1) | 1 (1)
Spinal cord infarction (Nervous system disorders) | 1 (1) | 0 (0)
Spinal cord oedema (Nervous system disorders) | 0 (0) | 1 (1)
Status epilepticus (Nervous system disorders) | 1 (1) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 4 (4) | 4 (4)
Syncope (Nervous system disorders) | 46 (48) | 52 (54)
Thalamus haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Thrombotic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Toxic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Transient global amnesia (Nervous system disorders) | 0 (0) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 37 (44) | 39 (42)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Trigeminal neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Uraemic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Vascular dementia (Nervous system disorders) | 0 (0) | 1 (1)
Vascular encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Vasogenic cerebral oedema (Nervous system disorders) | 0 (0) | 1 (1)
Vertebral artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Vertebrobasilar insufficiency (Nervous system disorders) | 2 (2) | 1 (1)
Vertigo cns origin (Nervous system disorders) | 0 (0) | 1 (1)
Viith nerve paralysis (Nervous system disorders) | 2 (2) | 3 (3)
Vith nerve paralysis (Nervous system disorders) | 1 (1) | 1 (1)
Vith nerve paresis (Nervous system disorders) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1/1394 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1/1394 (1)
Abnormal behaviour (Psychiatric disorders) | 1 (1) | 0 (0)
Acute psychosis (Psychiatric disorders) | 0 (0) | 1 (1)
Acute stress disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Adjustment disorder (Psychiatric disorders) | 1 (1) | 1 (1)
Adjustment disorder with anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Adjustment disorder with depressed mood (Psychiatric disorders) | 1 (1) | 0 (0)
Adjustment disorder with mixed disturbance of emotion and conduct (Psychiatric disorders) | 1 (1) | 0 (0)
Aggression (Psychiatric disorders) | 1 (1) | 1 (1)
Alcohol abuse (Psychiatric disorders) | 2 (2) | 4 (4)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1) | 1 (1)
Alcoholism (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (3) | 2 (3)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 2 (2) | 1 (1)
Confusional state (Psychiatric disorders) | 3 (3) | 5 (5)
Delirium (Psychiatric disorders) | 2 (2) | 3 (3)
Delirium tremens (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 4 (4) | 2 (2)
Depression suicidal (Psychiatric disorders) | 0 (0) | 1 (1)
Generalised anxiety disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1)
Hypomania (Psychiatric disorders) | 0 (0) | 1 (2)
Major depression (Psychiatric disorders) | 2 (3) | 1 (1)
Mental disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 3 (3) | 13 (15)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1)
Post-traumatic stress disorder (Psychiatric disorders) | 1 (3) | 0 (0)
Psychogenic seizure (Psychiatric disorders) | 1 (1) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 2 (2)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 48 (58) | 67 (81)
Acute prerenal failure (Renal and urinary disorders) | 0 (0) | 2 (2)
Azotaemia (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder outlet obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder prolapse (Renal and urinary disorders) | 0 (0) | 2 (2)
Calculus ureteric (Renal and urinary disorders) | 7 (7) | 9 (9)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 9 (10) | 10 (11)
Cystitis haemorrhagic (Renal and urinary disorders) | 0 (0) | 1 (1)
Cystitis ulcerative (Renal and urinary disorders) | 0 (0) | 1 (1)
Diabetic nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Glomerulonephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Glomerulosclerosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 11 (14) | 4 (4)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 5 (5)
Hypotonic urinary bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 19 (20) | 10 (12)
Nephropathy (Renal and urinary disorders) | 2 (2) | 0 (0)
Nephrosclerosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 2 (2)
Obstructive uropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Pelvi-ureteric obstruction (Renal and urinary disorders) | 0 (0) | 1 (2)
Prerenal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 3 (3) | 5 (5)
Renal colic (Renal and urinary disorders) | 2 (2) | 2 (2)
Renal cyst (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 14 (16) | 11 (11)
Renal haematoma (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 3 (3) | 2 (2)
Renal infarct (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1) | 2 (2)
Renal vein thrombosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Stress urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureteral disorder (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 2 (2) | 3 (3)
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 4 (4) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (2) | 9 (9)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Amastia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 10/4648 (10) | 12/4658 (12)
Cervical polyp (Reproductive system and breast disorders) | 0 (0) | 1/1394 (1)
Cystocele (Reproductive system and breast disorders) | 1/1388 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1/1394 (1)
Menometrorrhagia (Reproductive system and breast disorders) | 0 (0) | 1/1394 (1)
Ovarian cyst (Reproductive system and breast disorders) | 2/1388 (2) | 1/1394 (1)
Penile necrosis (Reproductive system and breast disorders) | 0 (0) | 1/4658 (1)
Peyronie's disease (Reproductive system and breast disorders) | 1/4648 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 4/4648 (5) | 2/4658 (2)
Rectocele (Reproductive system and breast disorders) | 0 (0) | 1/1394 (1)
Testicular disorder (Reproductive system and breast disorders) | 1/4648 (1) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 1/1388 (1) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 2/1388 (2) | 2/1394 (2)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 5 (5)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 14 (16) | 20 (20)
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 5 (7)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 43 (55) | 47 (55)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 26 (29) | 23 (23)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 10 (10)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 6 (6)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 7 (11)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 4 (4)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Mediastinal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pickwickian syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 12 (13)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 8 (11)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (3)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 21 (22) | 20 (20)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (5)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 8 (8)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 17 (17) | 16 (17)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Tracheomalacia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Dermatomyositis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 10 (11) | 3 (4)
Diabetic neuropathic ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Henoch-schonlein purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 9 (9) | 5 (6)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Vasculitic rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Abdominal hernia repair (Surgical and medical procedures) | 1 (1) | 2 (2)
Adrenalectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Amputation (Surgical and medical procedures) | 0 (0) | 1 (2)
Analgesic therapy (Surgical and medical procedures) | 1 (1) | 0 (0)
Aneurysm repair (Surgical and medical procedures) | 1 (1) | 1 (1)
Angioplasty (Surgical and medical procedures) | 12 (12) | 8 (9)
Ankle arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Aortic aneurysm repair (Surgical and medical procedures) | 4 (4) | 1 (1)
Aortic bypass (Surgical and medical procedures) | 1 (1) | 1 (1)
Aortic valve repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Aortic valve replacement (Surgical and medical procedures) | 4 (4) | 1 (1)
Arterial stent insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Atherectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Atrial septal defect repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Autonomic nerve operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Bladder neck suspension (Surgical and medical procedures) | 1/1388 (1) | 0 (0)
Bone operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Bronchial lesion excision (Surgical and medical procedures) | 0 (0) | 1 (1)
Cancer surgery (Surgical and medical procedures) | 1 (1) | 1 (1)
Cardiac ablation (Surgical and medical procedures) | 3 (5) | 6 (6)
Cardiac pacemaker battery replacement (Surgical and medical procedures) | 1 (1) | 3 (3)
Cardiac pacemaker insertion (Surgical and medical procedures) | 6 (6) | 3 (4)
Cardiac pacemaker replacement (Surgical and medical procedures) | 1 (1) | 1 (1)
Cardiac rehabilitation therapy (Surgical and medical procedures) | 1 (1) | 3 (4)
Cardiac resynchronisation therapy (Surgical and medical procedures) | 0 (0) | 2 (2)
Cardioversion (Surgical and medical procedures) | 0 (0) | 1 (1)
Carotid angioplasty (Surgical and medical procedures) | 1 (1) | 1 (1)
Carotid endarterectomy (Surgical and medical procedures) | 3 (3) | 6 (6)
Carotid revascularisation (Surgical and medical procedures) | 1 (1) | 2 (2)
Carpal tunnel decompression (Surgical and medical procedures) | 1 (1) | 1 (1)
Cataract operation (Surgical and medical procedures) | 3 (4) | 4 (5)
Catheter placement (Surgical and medical procedures) | 0 (0) | 1 (1)
Cholecystectomy (Surgical and medical procedures) | 2 (2) | 5 (5)
Colectomy (Surgical and medical procedures) | 4 (4) | 1 (1)
Colostomy closure (Surgical and medical procedures) | 2 (2) | 1 (1)
Coronary angioplasty (Surgical and medical procedures) | 13 (16) | 21 (23)
Coronary arterial stent insertion (Surgical and medical procedures) | 11 (11) | 12 (13)
Coronary artery bypass (Surgical and medical procedures) | 54 (54) | 59 (59)
Coronary revascularisation (Surgical and medical procedures) | 82 (92) | 79 (89)
Cox-maze procedure (Surgical and medical procedures) | 1 (1) | 0 (0)
Debridement (Surgical and medical procedures) | 0 (0) | 1 (1)
Diaphragmatic operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Elective surgery (Surgical and medical procedures) | 1 (2) | 0 (0)
Endarterectomy (Surgical and medical procedures) | 2 (2) | 2 (2)
Endovenous ablation (Surgical and medical procedures) | 1 (1) | 0 (0)
Explorative laparotomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Exploratory operation (Surgical and medical procedures) | 1 (1) | 1 (1)
Eye operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Foot amputation (Surgical and medical procedures) | 1 (1) | 0 (0)
Gastrectomy (Surgical and medical procedures) | 1 (1) | 2 (2)
Gastric bypass (Surgical and medical procedures) | 2 (2) | 1 (1)
Gastrointestinal endoscopic therapy (Surgical and medical procedures) | 0 (0) | 2 (2)
Haematoma evacuation (Surgical and medical procedures) | 1 (1) | 0 (0)
Heart valve replacement (Surgical and medical procedures) | 0 (0) | 2 (2)
Hernia repair (Surgical and medical procedures) | 1 (1) | 3 (3)
High frequency ablation (Surgical and medical procedures) | 0 (0) | 1 (1)
Hip arthroplasty (Surgical and medical procedures) | 11 (12) | 7 (7)
Hip surgery (Surgical and medical procedures) | 1 (1) | 1 (1)
Hospitalisation (Surgical and medical procedures) | 1 (1) | 0 (0)
Hysterectomy (Surgical and medical procedures) | 1/1388 (1) | 1/1394 (1)
Implantable defibrillator insertion (Surgical and medical procedures) | 11 (11) | 13 (13)
Implantable defibrillator replacement (Surgical and medical procedures) | 1 (1) | 1 (1)
Incisional drainage (Surgical and medical procedures) | 1 (1) | 0 (0)
Incisional hernia repair (Surgical and medical procedures) | 2 (2) | 0 (0)
Inguinal hernia repair (Surgical and medical procedures) | 1 (1) | 5 (5)
Intervertebral disc operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Intraocular lens implant (Surgical and medical procedures) | 2 (3) | 1 (1)
Joint arthroplasty (Surgical and medical procedures) | 3 (3) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 12 (14) | 12 (12)
Knee operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Leg amputation (Surgical and medical procedures) | 5 (6) | 3 (3)
Lens extraction (Surgical and medical procedures) | 1 (2) | 1 (1)
Lipoma excision (Surgical and medical procedures) | 0 (0) | 1 (1)
Mastectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Medical device change (Surgical and medical procedures) | 1 (1) | 0 (0)
Medical device removal (Surgical and medical procedures) | 3 (3) | 0 (0)
Mitral valve replacement (Surgical and medical procedures) | 2 (2) | 0 (0)
Nephrectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Open reduction of fracture (Surgical and medical procedures) | 1 (1) | 0 (0)
Osteosynthesis (Surgical and medical procedures) | 0 (0) | 1 (1)
Osteotomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Pancreatectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Pancreaticoduodenectomy (Surgical and medical procedures) | 0 (0) | 2 (2)
Penile repair (Surgical and medical procedures) | 0 (0) | 1/4658 (1)
Percutaneous coronary intervention (Surgical and medical procedures) | 192 (217) | 182 (214)
Peripheral artery angioplasty (Surgical and medical procedures) | 3 (5) | 4 (5)
Peripheral artery bypass (Surgical and medical procedures) | 5 (5) | 6 (6)
Peripheral artery stent insertion (Surgical and medical procedures) | 0 (0) | 2 (3)
Peripheral endarterectomy (Surgical and medical procedures) | 3 (3) | 6 (6)
Peripheral nerve transposition (Surgical and medical procedures) | 0 (0) | 1 (1)
Peripheral revascularisation (Surgical and medical procedures) | 2 (2) | 2 (2)
Prostate ablation (Surgical and medical procedures) | 0 (0) | 1 (1)
Prostatectomy (Surgical and medical procedures) | 0 (0) | 2/4658 (2)
Radioactive iodine therapy (Surgical and medical procedures) | 1 (1) | 0 (0)
Rectal prolapse repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Renal artery angioplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Renal sympathetic nerve ablation (Surgical and medical procedures) | 0 (0) | 2 (2)
Resection of rectum (Surgical and medical procedures) | 1 (1) | 1 (1)
Resuscitation (Surgical and medical procedures) | 0 (0) | 1 (1)
Retinopexy (Surgical and medical procedures) | 0 (0) | 1 (1)
Rotator cuff repair (Surgical and medical procedures) | 1 (1) | 1 (1)
Shoulder arthroplasty (Surgical and medical procedures) | 2 (2) | 0 (0)
Shoulder operation (Surgical and medical procedures) | 1 (1) | 1 (1)
Skin neoplasm excision (Surgical and medical procedures) | 1 (2) | 1 (1)
Spinal decompression (Surgical and medical procedures) | 1 (1) | 1 (1)
Spinal fusion surgery (Surgical and medical procedures) | 5 (5) | 1 (1)
Spinal laminectomy (Surgical and medical procedures) | 4 (4) | 3 (3)
Spinal operation (Surgical and medical procedures) | 1 (1) | 1 (1)
Stent placement (Surgical and medical procedures) | 3 (3) | 2 (2)
Sympathectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Tenotomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Therapeutic embolisation (Surgical and medical procedures) | 1 (1) | 0 (0)
Therapy cessation (Surgical and medical procedures) | 0 (0) | 1 (1)
Thrombectomy (Surgical and medical procedures) | 3 (3) | 1 (1)
Thrombosis prophylaxis (Surgical and medical procedures) | 1 (1) | 1 (1)
Thyroidectomy (Surgical and medical procedures) | 3 (3) | 0 (0)
Toe amputation (Surgical and medical procedures) | 1 (1) | 4 (4)
Tongue operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Total adrenalectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Transmyocardial revascularisation (Surgical and medical procedures) | 2 (2) | 0 (0)
Transurethral bladder resection (Surgical and medical procedures) | 0 (0) | 1 (1)
Transurethral prostatectomy (Surgical and medical procedures) | 2/4648 (2) | 1/4658 (1)
Tricuspid valve repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Tumour excision (Surgical and medical procedures) | 0 (0) | 1 (1)
Ureteral stent insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Ureteral stent removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Vaginal prolapse repair (Surgical and medical procedures) | 1/1388 (1) | 0 (0)
Valvuloplasty cardiac (Surgical and medical procedures) | 1 (1) | 0 (0)
Vascular graft (Surgical and medical procedures) | 0 (0) | 1 (1)
Venous stent insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Ventricular assist device insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Vitrectomy (Surgical and medical procedures) | 0 (0) | 2 (2)
Wound drainage (Surgical and medical procedures) | 1 (1) | 0 (0)
Accelerated hypertension (Vascular disorders) | 2 (2) | 1 (1)
Aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 18 (18) | 14 (14)
Aortic aneurysm rupture (Vascular disorders) | 3 (3) | 1 (1)
Aortic dissection (Vascular disorders) | 0 (0) | 1 (1)
Aortic elongation (Vascular disorders) | 0 (0) | 1 (1)
Aortic occlusion (Vascular disorders) | 0 (0) | 1 (1)
Aortic rupture (Vascular disorders) | 0 (0) | 2 (2)
Aortic stenosis (Vascular disorders) | 18 (18) | 17 (19)
Aortitis (Vascular disorders) | 1 (1) | 0 (0)
Arterial disorder (Vascular disorders) | 1 (1) | 0 (0)
Arterial haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Arterial insufficiency (Vascular disorders) | 1 (1) | 1 (1)
Arterial occlusive disease (Vascular disorders) | 3 (4) | 1 (1)
Arterial perforation (Vascular disorders) | 1 (1) | 0 (0)
Arterial stenosis (Vascular disorders) | 1 (1) | 0 (0)
Arterial thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (1) | 3 (3)
Artery dissection (Vascular disorders) | 1 (1) | 0 (0)
Axillary vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Blood pressure inadequately controlled (Vascular disorders) | 1 (1) | 0 (0)
Brachiocephalic artery stenosis (Vascular disorders) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 1 (1) | 3 (3)
Deep vein thrombosis (Vascular disorders) | 11 (12) | 16 (16)
Dry gangrene (Vascular disorders) | 0 (0) | 2 (3)
Embolism arterial (Vascular disorders) | 1 (1) | 0 (0)
Extremity necrosis (Vascular disorders) | 1 (1) | 1 (1)
Femoral artery aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Femoral artery occlusion (Vascular disorders) | 7 (8) | 7 (7)
Femoral artery perforation (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 7 (7) | 3 (3)
Haemorrhage (Vascular disorders) | 0 (0) | 3 (3)
Hypertension (Vascular disorders) | 21 (23) | 18 (19)
Hypertensive crisis (Vascular disorders) | 9 (9) | 14 (16)
Hypertensive emergency (Vascular disorders) | 3 (3) | 0 (0)
Hypotension (Vascular disorders) | 11 (12) | 17 (18)
Hypovolaemic shock (Vascular disorders) | 2 (2) | 1 (1)
Iliac artery occlusion (Vascular disorders) | 2 (2) | 3 (3)
Iliac artery rupture (Vascular disorders) | 1 (1) | 0 (0)
Intermittent claudication (Vascular disorders) | 7 (7) | 16 (20)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 2 (2)
Lymphatic fistula (Vascular disorders) | 0 (0) | 1 (1)
Lymphorrhoea (Vascular disorders) | 0 (0) | 1 (1)
Malignant hypertension (Vascular disorders) | 4 (4) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 11 (11) | 4 (4)
Peripheral arterial occlusive disease (Vascular disorders) | 52 (66) | 50 (66)
Peripheral artery aneurysm (Vascular disorders) | 2 (2) | 2 (2)
Peripheral artery stenosis (Vascular disorders) | 19 (21) | 10 (10)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 6 (7)
Peripheral embolism (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 12 (14) | 20 (25)
Peripheral vascular disorder (Vascular disorders) | 21 (25) | 10 (11)
Shock (Vascular disorders) | 0 (0) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 1 (1)
Subclavian artery occlusion (Vascular disorders) | 0 (0) | 2 (2)
Subclavian artery stenosis (Vascular disorders) | 2 (3) | 4 (4)
Subclavian artery thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Temporal arteritis (Vascular disorders) | 2 (2) | 0 (0)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 2 (2) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Varicose vein (Vascular disorders) | 2 (2) | 2 (2)
Vascular occlusion (Vascular disorders) | 2 (2) | 0 (0)
Vasculitis (Vascular disorders) | 0 (0) | 1 (1)
Vena cava thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Evacetrapib (N=6036) | Placebo (N=6052)
Diarrhoea (Gastrointestinal disorders) | 472 (568) | 414 (484)
Bronchitis (Infections and infestations) | 363 (456) | 375 (443)
Nasopharyngitis (Infections and infestations) | 452 (603) | 465 (602)
Upper respiratory tract infection (Infections and infestations) | 327 (397) | 327 (410)
Arthralgia (Musculoskeletal and connective tissue disorders) | 375 (426) | 370 (425)
Back pain (Musculoskeletal and connective tissue disorders) | 399 (442) | 379 (412)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 339 (412) | 329 (388)
Dizziness (Nervous system disorders) | 389 (435) | 352 (407)
Cough (Respiratory, thoracic and mediastinal disorders) | 327 (367) | 279 (304)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 305 (339) | 307 (341)
Hypertension (Vascular disorders) | 453 (508) | 403 (466)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days